CLINICAL TRIAL: NCT04428749
Title: Swallowing Difficulties in ICU Patients [Synkebesvær Hos Intensivpatienter]
Acronym: ICU-Swallow
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospitalsenheden Vest (Other)
Collaborators: VIA University College (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Anne Højager Nielsen, Principal Investigator, MCN, PH.D., Hospitalsenheden Vest
Other Study IDs: 69184
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Deglutition Disorders; Critical Illness
MeSH Terms: conditions — Deglutition Disorders; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: 1. Participants are screened using the Yale Swallow Protocol (YSP) 2-4 hours after extubation:
     Ability to swallow is assessed by an ICU nurse using the YSP. If the YSP is negative, the patient may start oral feeding and drinking. In case of a positive YSP, the screening may be repeated within the next 24 hours provided the patient improves clinically. If YSP continues to be positive the patient is referred to assessment by a speech language pathologist (SLP).
  2. Participants are screened within 24 hours:
  To evaluate YSP against the FEES, the patient undergoes 1) YSP performed by an ICU nurse followed by 2) FEES performed by a SLP (until PAS>6 (aspiration on any food consistency on the Penetration Aspiration Scale (20)). The SLP will be blinded to the assessment made by the ICU nurses. Patients will follow recommendations for oral feeding and drinking as given by the SLP.
  Interventions: Diagnostic Test: Yale Swallow Protocol; Diagnostic Test: FEES (fiberoptic endoscopic evaluation of swallowing)

INTERVENTIONS:
Diagnostic Test: Yale Swallow Protocol — The YSP is a three-step method consisting of an assessment of the patient's awareness, the patient's ability to follow simple instructions and finally the patient's ability to drink 90 ml water from a cup or by straw without stopping, choking or coughing.
Diagnostic Test: FEES (fiberoptic endoscopic evaluation of swallowing) — The FEES will be performed bedside by an experienced occupational therapists. The patient will be sitting upright in a chair and be given 1) 2 spoons of applesauce, 2) 2 spoons of water, 3) several sips of water, 4) 90 ml of water. All items colored blue.
  The FEES will use a single-use AMBU rhino-laryngo scope slim and the AMBU monitor. the examination will be terminated in case of aspiration below the vocal cords.

SUMMARY:
Swallow disorders or dysphagia related to mechanical ventilation affects between 1,300 and 2,000 patients in Danish intensive care units every year and increases aspiration, pneumonia and risk of dying. In intensive care units, dysphagia may vary around the clock as fatigue and fluctuating alertness play an important role for the patients' ability to swallow effectively without aspiration to the airway. For this reason, ICU nurses must be able to assess dysphagia in the ICU patient day and night, but guidelines are lacking.

One of the simplest and most sensitive methods is the Yale Swallow Protocol, however, this protocol requires translation and validation before it can be implemented in Danish intensive care units. This project aims to translate and validate the Yale Swallow Protocol for use in Danish intensive care units. Furthermore, this project will explore nurses' perceptions and management of dysphagia in the intensive care unit as well as feasibility and acceptability of the Yale Swallow Protocol.

DETAILED DESCRIPTION:
Introduction Dysphagia caused by intubation and mechanical ventilation affects between 1.300 - 2.000 patients in Danish intensive care units (ICU's) every year. Dysphagia increases the risk of aspiration, pneumonia, repeated mechanical ventilation and mortality. Despite this, national and international guidelines for treating dysphagia in the ICU are lacking. In ICU patients, dysphagia may vary around the clock as fatigue and cerebral status plays an important role for the patients' ability to swallow effectively without aspiration. For this reason, ICU nurses must be able to assess dysphagia in the ICU patient day and night. This will be an important addition to assessments made by occupational therapists usually only available in the morning hours. However, for nurses to be able to assess dysphagia in the ICU patients; development and validation of screening procedures are highly needed.

The development of a validated screening procedure to detect dysphagia in ICU patients will furthermore pave the way for the developing and testing nursing interventions aiming at improving dysphagia in ICU patients. This may reduce complications and improve quality of life in patients.

Dysphagia related to mechanical ventilation and intensive care The swallow function depends on a complicated interplay between more than 30 muscle pairs, cranial nerves and areas in the cortex and the medulla oblongata. Causes for dysphagia in ICU patients are only partially understood, however, the following factors have been suggested as significant: 1) Trauma to the pharynx caused by intubation (placing a tube for mechanical ventilation in the airway), 2) Neuromyopathy resulting in muscular weakness, 3) Decreased level of consciousness caused by medication, delirium or critical illness. Moreover, these factors may cause dysphagia in ICU patients to vary from day to night.

Dysphagia is a serious complication to critical illness, potentially increasing mortality. Despite this, research shows that nursing practice varies greatly. Nurses have different views on what constitutes safe swallowing. Nonetheless, it often falls upon nurses to assess patients swallowing function and determine whether to offer the patient something to eat and drink or not. Thus, developing valid screening methods that can be used by ICU nurses may improve patient safety and reduce complications due to dysphagia caused by intubation, mechanical ventilation and critical illness.

Diagnosing dysphagia using FEES Dysphagia can be diagnosed using instrumental methods such as the fiberoptic endoscopic evaluation of swallowing (FEES). This method is considered a gold standard in assessing dysphagia. FEES may be performed bed-side by physicians or occupational therapists by testing different foods and consistencies, but some patients find the FEES disagreeable. A clinical examination by occupational therapists is another way to diagnose dysphagia, however, silent aspiration without choking or coughing is difficult to detect in a clinical examination.

(NOTE: In Denmark, the speech language therapist is usually an occupational therapist).

Screening for dysphagia Screening for dysphagia in general hospital populations is possible by using different screening methods.

One of the most rigorously validated tests is the Yale Swallow Protocol (YSP). The YSP is a three-step method consisting of an assessment of the patient's awareness, the patient's ability to follow simple instructions and finally the patient's ability to drink 90 ml water from a cup or by straw without stopping, choking or coughing. The YSP has high sensitivity of 0.96, thus effectively identifying patients who may safely begin oral feeding and drinking. The specificity 0.5 indicates that patients who fail the YSP will need a specialized assessment before eating and drinking is commenced. The clinical importance of this is that nurses may employ the YSP at all hours to identify patients at risk, and thereby be able to prevent aspiration detrimental to patient recovery. Moreover, patients not at risk can begin oral feeding earlier, which may improve nutritional status and wellbeing in the patient. However, dysphagia in ICU patients varies from other hospital patients because of intubation, muscle weakness and alternating level of consciousness. Therefore it is necessary to validate a translated version of the YSP on ICU patients to determine its predictive abilities. In addition, skilled clinicians' uptake of a new screening method is a complex process. Therefore, the feasibility and acceptability of the YSP in a Danish ICU needs to be explored before the YSP can be recommended for implementation on a greater scale.

Research questions

1. Is systematic screening of dysphagia in ICU patients using the Yale Swallow protocol feasible and acceptable to clinicians and patients?
2. Can the Yale Swallow Protocol, administered by ICU nurses bed side 24 hours a day, identify dysphagia in ICU patients? What are the predictive abilities compared to FEES (gold standard)?

Methods

STUDY 1

Design: Feasibility study. The aim of this study is to explore feasibility of implementing and evaluating the YSP in a regional ICU and acceptability among clinicians and patients. This includes exploring barriers and facilitators to screening ICU patients for dysphagia, fidelity to the YSP and FEES methods and fidelity to recommendations for oral intake of food and drinks based on the YSP and FEES.

The four-phased feasibility study will address feasibility of both the YSP and research methods for study 2.

STUDY 2

Design: Prospective observational study, which will be adjusted based on the feasibility study (study 1).

Intervention:

A. Screening 2-4 hours after extubation:

Ability to swallow is assessed by an ICU nurse using the YSP. If the YSP is negative, the patient may start oral feeding and drinking. In case of a positive YSP, the screening may be repeated within the next 24 hours provided the patient improves clinically. If YSP continues to be positive the patient is referred to assessment by a speech language pathologist (SLP).

B. Screening within 24 hours:

To evaluate YSP against the FEES, the patient undergoes 1) YSP performed by an ICU nurse followed by 2) FEES performed by an occupational therapist (until PAS>6 (aspiration on any food consistency on the Penetration Aspiration Scale). The occupational therapist will be blinded to the assessment made by the ICU nurses. Patients will follow recommendations for oral feeding and drinking as given by the occupational therapist.

Data:

For patients, the following data will be recorded: time and results of the initial YSP screening 2-4 hours post extubation, recommendation for oral feeding and drinking, time and results of the YSP and the FEES performed within 24 hours of extubation and recommendation for oral feeding and drinking. In addition, sex, age, diagnosis, Simplified Acute Physiology Score (SAPSIII) , Charlson Comorbidity Index, chronic obstructive pulmonary disease, length of stay in hospital, length of stay in ICU, time on mechanical ventilation, new pneumonia following extubation, FOIS (Functional Oral Intake Scale) and death within 30 days.

For clinicians performing the YSP and FEES, the following data will be recorded: age, sex, profession, experience in years, and ICU experience in years.

Sample size: Given a prevalence of dysphagia among acute ICU patients of 18 %; a sensitivity of YSP of 0.96 and a specificity of 0.5, then inclusion of 25 patients will be able to show a negative likelihood ratio (LR-) of 0.1 [95 % CI 0,00; 5,74], which means that almost all patients passing the YSP will be without dysphagia. Estimating the attrition rate to be 25 %, 35 patients will be included in the study.

Analysis: Screening by YSP and assessment by FEES with 24 hours will be tabulated in a 2x2 table, calculating the sensitivity, specificity, positive predictive value and negative predictive value of YSP compared to FEES. Correlations between patient characteristics will be calculated using Pearson and Spearman correlation statistics as appropriate.

Research ethics

All participants receive written and oral information about the purpose of the study and give signed, informed consent. Relatives of patients are informed about the study. In case a participant is affected adversely by participation, support will be offered by nurses and physicians from the ICU.

The study is approved by the Health Research Committee of Region Central Jutland. The study is registered with Danish Data protection Agency and data will be stored in REDCap hosted by Aarhus University and Midt-X, a research data site hosted by the Central Denmark Region.

All data will be anonymized before shared or published; all data will be published.

Perspectives

If screening with the YSP can identify dysphagia in the critically ill patients, this will allow oral feeding and drinking in many patients, leading to improved nutritional status and increased patient satisfaction with no compromise of patient safety. Moreover, an effective screening method for dysphagia may pave the way for developing nursing interventions to prevent dysphagia from developing in the intensive care patient. In turn, this may reduce complications, human suffering and costs.

ELIGIBILITY:
Inclusion criteria:

* > 18 years
* No prior records of dysphagia
* Extubated after mechanical ventilation > 24 hours.
* Awake and alert with no sign of ICU delirium.
* Must understand Danish, as all information available about the study is in Danish.

Exclusion criteria:

* Patients who are unable to undergo the YSP
* Patients who are unable to undergo the FEES

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients from all clinical specialties who have been extubated after mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-12 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Aspiration on FEES | Within 24 hours of extubation
  Penetration aspiration scale (PAS scale) equal to or larger than 6
Yale Swallow protocol | Within 30 minutes of the FEES
  Passed or not passed

SECONDARY OUTCOMES:
Mortality | 30 days after extubation
  Dead or alive according to patient record

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Nielsen, Ph.d., Principal Investigator — Regional Hospital Holstebro
Locations (1):
- Regionshospitalet Holstebro, Holstebro, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided